CLINICAL TRIAL: NCT00562666
Title: Immunotherapy of Hepatocellular Carcinoma by Hepatic Intra Arterial Injection of Autologous Gamma-delta T Lymphocytes: A Phase I Study
Brief Title: Immunotherapy of Hepatocellular Carcinoma With Gamma Delta T Cells
Acronym: ICAR
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID RCB 2007-A00249-44; CIC 0203/074; LOC 06/07
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: cell therapy; T lymphocytes; hepatic intra-arterial injection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Single hepatic intra arterial administration of 500 millions T gamma delta lymphocytes
  Interventions: Other: T gamma delta lymphocytes
- 2 (Experimental): Single hepatic intra arterial administration of 1000 millions T gamma delta lymphocytes
  Interventions: Other: T gamma delta lymphocytes
- 3 (Experimental): Single hepatic intra arterial administration of 2000 millions T gamma delta lymphocytes
  Interventions: Other: T gamma delta lymphocytes
- 4 (Experimental): Single hepatic intra arterial administration of 4000 millions T gamma delta lymphocytes
  Interventions: Other: T gamma delta lymphocytes

INTERVENTIONS:
Other: T gamma delta lymphocytes — Single hepatic intra arterial administration of increasing doses of T gamma delta lymphocytes

SUMMARY:
For most patients with hepatocellular carcinoma, surgery or other curative procedures are not possible and only palliative measures could be applied (chemoembolization, targeted drugs, best supportive cares, etc). In the ICAR study, increasing doses of a cell therapy product will be evaluated in patients in a palliative setting. All patients will have one hepatic intra-arterial injection of immunological cells (gamma-delta T lymphocytes) and will be evaluated for safety.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18
* Hepatocellular carcinoma histologically proven, with at least one measurable tumor
* Non operable tumor
* Alfa foeto protein > 400 ng/ml
* Other treatments (surgery, chemoembolization) non indicated
* Chemoembolization non indicated due to good performance status (WHO 1) or to tumor volume
* Performance status WHO < 2
* Life expectancy > 3 months

Non inclusion Criteria:

* Extra hepatic metastases
* Severe hepatopathy (Child B or C)
* Virus B or C chronic hepatitis
* Chronic cardiac failure
* Uncontrolled severe infectious disease
* Other cancer, if not considered as cured
* Positive serology for HIV or HTLV
* Leucocytes < 3000/mm3 or neutrophils < 1500/mm3
* Platelets < 80000/mm3
* Serum creatinine > 110 µmol/L
* Bilirubin > 35 µmol/L
* AST, ALT, alkaline phosphatase > 5N
* Current immunosuppressive treatment
* Impossibility to comply with scheduled follow-up
* Anatomical situation not permitting the selective injection of the product of cell therapy
* Pregnant or breastfeeding woman, or not using adequate effective contraceptive method

Exclusion Criterion:

* Insufficient number of gamma delta lymphocytes after expansion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Onset of: thrombosis of hepatic artery, grade 4 liver toxicity, or grade 3 or more allergic, neurological, dermatological, infectious, or respiratory reaction | Within 14 days after treatment

SECONDARY OUTCOMES:
Onset of clinical, biological signs or images evocative of lymphocyte-induced tumor cytotoxicity and/or of a persistence of gamma-delta T cells in peripheral blood. Tumor response will be evaluated with the RECIST criteria. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc RAOUL, MD, PhD, Principal Investigator — CRLCC Eugène Marquis, Rennes; Eric BELLISSANT, MD, PhD, Study Chair — Rennes University Hospital
Locations (3):
- France (3):
  - Unité de Thérapie Cellulaire, Laboratoire de Cytogénétique et Biologie Cellulaire, CHU Rennes, Rennes
  - Département d'Oncologie Médicale - CRLCC Eugène Marquis, Rennes
  - Service de Chirugie Viscérale - Hôpital de Pontchaillou, Rennes